CLINICAL TRIAL: NCT05052047
Title: Effects of 30 Min Brisk Walk on HRLQ and Pulmonary Functions on COPD Patients
Brief Title: Brisk Walk on Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01081 Shiza Zafar
Record Dates: First submitted 2021-09-18; First posted 2021-09-22 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: COPD
Keywords: Aerobic Exercise; Brisk Walk; Health-related quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brisk Walking Group (Experimental): Brisk walking as training for 4 weeks
  Interventions: Other: Brisk Walking Group
- Conventional Breathing Exercise Group (Active Comparator): Conventional Breathing exercise for 4 weeks
  Interventions: Other: Conventional Breathing Exercise Group

INTERVENTIONS:
Other: Brisk Walking Group — Brisk Walk: 20 min/day (The researchers found, for most people, brisk walking could be defined as moving at a pace of 2.7 miles per hour or 100 steps per minute for adults under about age 60 or guidelines define brisk walking as occurring when individuals move at a pace that increases their heart rate to about 70% of their heart rate maximum) Patient will also perform breathing exercises as given to Control group, Positioning (lean forward when needed) Percussion coughing when needed
  Arms: Brisk Walking Group
Other: Conventional Breathing Exercise Group — Breathing exercises: 20 min/day
  Breathing Ex includes:
  • Pursed lip breathing: Sit with your back straight, inhale through your nose for 2 seconds. Purse your lips like you rae blowing on hot food and then breath out slowly, take twice as long to exhale as you took to breath in 4-5 times a day
  • Diaphragmatic breathing: Lie on your back on a flat surface, knees bent and head supported. Use pillow under knees to support your legs . breathe in slowly through your nose tighten your stomach, letting them fall inward as you exhale through your pursed lips. Practice these exercises 5-10 minutes about 3-4 times a day.
  Positioning (lean forward when needed) Percussion coughing when needed
  Arms: Conventional Breathing Exercise Group

SUMMARY:
To determine the effects of 30 min brisk walk on Pulmonary Functions on COPD patients To determine the effects of 30 min brisk walk on Health related Health-related quality of life (HRLQ) on Chronic obstructive pulmonary disease (COPD) patients

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (GOLD criteria Mild and Moderate).

Exclusion Criteria:

* Dyspnea more than 4
* Walking issues
* Rheumatoid arthritis
* Musculoskeletal disorder
* Acute infections.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
6 min walk test: Distance (meters) | 4th Week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Peak VO2max with formula | 4th Week
  Changes from the baseline, Maximal oxygen uptake or capacity is the maximum rate of oxygen consumed and measured during the stress activity. Its measurement within the laboratory demonstrates a numerical value for endurance fitness full stop and this value can be used to compare individuals training with or without diseases. This tool reflects cardiopulmonary endurance in the performance of any exercise. maximal oxygen consumption (VO2 max) is calculated by:
  Mean Peak VO2 (ml/kg/Mean) = 4.948 + 0.023 *Mean 6MWD (meters)
  6 minute walk distance (6MWD)
Health-related quality of life scale (HRLQ) | 4th week
  Changes from the baseline, It is usually administer the Health-Related Quality of Life scale verbally, reading the questions aloud and writing down respondents' answers.
  The scale consists of three modules. The Core Healthy Days module contains one item that asks respondents to rate their general health on a 5-point scale (1 = excellent; 3 = good; 5 = poor). The module also has three items that ask respondents how many days their physical health was not good, their mental health was not good, and their health interfered with their daily activities.
  It compute an unhealthy days score by adding the number of physically unhealthy and mentally unhealthy days. The maximum score is 30 unhealthy days, even if the number of unhealthy days totals more than 30.
Forced Expiratory Volume in 1 second (FEV1) | 4th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 4th week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 4th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

SECONDARY OUTCOMES:
Quality of life: St. George's Respiratory Questionnaire (SGRQ) | 4th week
  It is used to access the quality of life; SGRQ is used for determining quality of life in COPD patients. This questionnaire is designed in 50 items to check the impact of COPD. 0 to 100 is the range of this score. Scores having higher values means more limitations

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Capital Hospital Islamabad, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No